CLINICAL TRIAL: NCT05485324
Title: TREATMENT OF PAIN IN PATIENTS WITH Gunshot and Mine-explosive Wounds AT THE STAGES OF TREATMENT
Brief Title: The Concept of Pain Treatment in Patients With Gunshot and Mine-explosive Wounds and to Develop an Algorithm for Analgesia at the Stages of Treatment
Acronym: CPTGaM-EW
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Chief researcher, Bogomolets National Medical University
Other Study IDs: №158/23,05,2022
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
Keywords: concept of pain treatment, pain, wounds, stages of treatment
MeSH Terms: conditions — Chronic Pain; Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Interventions: Other: visual analog scale
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022
  Interventions: Other: visual analog scale

INTERVENTIONS:
Other: visual analog scale — Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Other Names: neuropathic pain Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36 (DN4).; Chaban Quality of Life Scale; The Hospital Anxiety and Depression Scale (HADS); Mississippi PTSD scale (military version)

SUMMARY:
in 82.1% of cases it is not possible to achieve a positive result of pain treatment

DETAILED DESCRIPTION:
The concept of pain treatment in patients with gunshot and mine-explosive injuries and the developed pain relief algorithm at the stages of treatment will have an impact on the results of pain treatment in this category of patients.

ELIGIBILITY:
Inclusion Criteria:

* the presence of gunshot and mine-explosive injuries

Exclusion Criteria:

* absence of gunshot and mine-explosive injuries

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
Sampling Method: Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  from 0 to 10 points
Didier Bouhassiraa DN4 | 12 months
  4 or more points (a neuropathic pain component is present)
The Hospital Anxiety and Depression Scale | 12 months
  0-7 is the norm 8-13 - mild depressive disorders 14-18 - depressive disorders of medium severity 19-22 - severe depressive disorders 23 and more - depressive disorders of a very severe degree of severity
Chaban Quality of Life Scale | 12 months
  up to 56 inclusive - a very low level 57-66 - low 67-75 - average 76-82 - tall 83-100 is very high
Mississippi PTSD scale (military version) | 12 months
  the mean values of the total score are 76±18 for well-adjusted servicemen, 86±26 for servicemen with mental disorders, and 130±18 for those with PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share